CLINICAL TRIAL: NCT02381587
Title: Retrospective Study That Evaluate the Effect of HCG Treatment as a Cardiovascular Disease Morbidity Factor in Patients With Primary Sjogren Syndrome
Brief Title: the Effect of HCG Treatment as a Cardiovascular Disease Morbidity Factor in Sjogren Syndrome Patients
Acronym: HAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yair levy, professor - head of internal medicine department, Meir Medical Center
Other Study IDs: HCQ and sjogren
Record Dates: First submitted 2015-02-16; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Primary Sjogren Syndrome With Multisystem Involvement
MeSH Terms: interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Retrospective study — no interventional study - Retrospective study that valuate The effect of HCQ treatment in cardiovascular AVENTS IN patients with primary sjogren syndrome

SUMMARY:
sjogren syndrome is an autoimmune disease that mainly affects the Salivary glands and Lacrimal gland In addition to the effects of this disease is characterized by overall systemic Muskals injury, pulmonary disease, peripheral neuropathy and vasculitis. In addition recent studies have shown that patients are at increased risk of the disease up to 2 cardiac events and stroke events Hydroxychloroquine is an RHEUMATIC DISEASE PROCESS SUPPRESSANTS-ANTIMALARIALS used to treat anti-inflammatory rheumatic diseases in many first-line treatment is sjogren syndrome.

A recent study of the treatment in Hydroxychloroquine effect on lipid profile sjogren syndrome patients showed a reduction in total cholesterol levels and increase in HDL. Further studies of the impact made Hydroxychloroquine systemic lupus patients erythematosus (SLE) showed in Atherosclerosis and morbidity and mortality reduction in cardiovascular. Studies of patients with rheumatoid arthritis (RA) demonstrated reduced risk of developing diabetes and improved lipid profile Research Goals valuate The effect of HCQ treatment in cardiovascular patients with primary sjogren syndrome

DETAILED DESCRIPTION:
Research Goals Valuate The effect of HCQ treatment in cardiovascular patients with primary sjogren syndrome Research Methods The study will included patients that diagnosed with sjogren syndrome and was treated in Meir Medical center during the years 2003-2014 During the study will collect information on confounding factors , Risk factors include cardiovascular acceptable such as diabetes, dyslipidemia, high blood pressure and the like, central nervous system involvement and steroid use

Study outcome will be one of the follow:

1. Thrombosis of peripheral veins
2. Arterial cardiovascular events
3. Cardiac events (myocardial infarction
4. Stroke (stroke and TIA)

4. Venous thrombosis events 5. Pulmonary embolism In the study will be 500 patients

Inclusion criteria:

1. 18 years old
2. Both sexes
3. Patients that diagnosis in sjogren in treated in Meir Medical center in the years 2003-2014 And treated in Hydroxychloroquine at least a month.

Exclusion criteria:

1. Minors and special populations
2. Patients that treated in Hydroxychloroquine at less than a month.
3. Patient that participate in clinical trial and treat with investigational product

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old
2. Both sexes
3. Patients that diagnosis in sjogren in treated in Meir Medical center in the years 2003-2014 And treated in Hydroxychloroquine at least a month.

Exclusion Criteria:

1. Minors and special populations
2. Patients that treated in Hydroxychloroquine at less than a month.
3. Patient that participate in clinical trial and treat with investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that diagnosis in sjogren in treated in Meir Medical center
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Arterial cardiovascular events | 15 years since the first dose of hydroxychloroquine

SECONDARY OUTCOMES:
Cardiac events (myocardial infarction | 15 years since the first dose of hydroxychloroquine
Thrombosis of peripheral veins | 15 years since the first dose of hydroxychloroquine
Stroke (stroke and TIA) | 15 years since the first dose of hydroxychloroquine
Venous thrombosis events | 15 years since the first dose of hydroxychloroquine
Pulmonary embolism | 15 years since the first dose of hydroxychloroquine